CLINICAL TRIAL: NCT02873702
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Dexlansoprazole (60 mg QD) and an Active Comparator, Lansoprazole (30 mg QD) on Healing of Erosive Esophagitis, and Maintenance of Healing in Subjects With Healed Erosive Esophagitis With Dexlansoprazole (30 mg QD) and Placebo
Brief Title: Efficacy and Safety of Dexlansoprazole in Healing and Maintaining Healing of Erosive Esophagitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Compound is not expected to change the current treatment practice or fill significant clinical need for patients in China over currently available EE agents.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-390MR_301; U1111-1142-0320 (Registry Identifier: WHO)
Record Dates: First submitted 2016-08-17; First posted 2016-08-19 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2018-10

CONDITIONS: Erosive Esophagitis
Keywords: Drug therapy
MeSH Terms: interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healing Period: Dexlansoprazole 60 mg (Experimental): Dexlansoprazole 60 milligram (mg), delayed-release capsules, orally, once daily for up to 8 weeks in the Healing Period.
  Interventions: Drug: Dexlansoprazole
- Healing Period: Lansoprazole 30 mg (Experimental): Lansoprazole 30 mg, capsules, orally, once daily for up to 8 weeks in the Healing Period.
  Interventions: Drug: Lansoprazole
- Maintenance Period: Dexlansprazole 30 mg (Experimental): Participants who will be healed at Week 8 will be randomized to receive dexlansoprazole 30 mg, delayed-release capsules, orally, once daily for up to 6 months in the Maintenance period.
  Interventions: Drug: Dexlansoprazole
- Maintenance Period: Placebo (Experimental): Participants who will be healed at Week 8 will be randomized to receive dexlansoprazole placebo-matching capsules, orally, once daily for up to 6 months in the Maintenance period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole delayed-release capsules.
  Arms: Healing Period: Dexlansoprazole 60 mg; Maintenance Period: Dexlansprazole 30 mg
Drug: Lansoprazole — Lansoprazole capsules.
  Arms: Healing Period: Lansoprazole 30 mg
Drug: Placebo — Dexlansoprazole placebo-matching capsules.
  Arms: Maintenance Period: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of dexlansoprazole compared to lansoprazole in healing erosive esophagitis (EE) in Chinese participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. Dexlansoprazole is being tested to treat people who have EE. This study will look at erosive esophageal healing in people who take dexlansoprazole.

The study will enroll approximately 450 participants. Participants will be randomly assigned to one of the two treatment groups with 1:1 ratio-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Dexlansoprazole 60 mg
* Lansoprazole 30 mg

After 8 weeks of treatment, participants will be evaluated to assess esophageal healing. If the EE is healed participants will be randomly assigned to one of two different treatment groups with 1:1 ratio:

* Dexlansoprazole 30 mg
* Placebo (dummy inactive pill) - this is a capsule that looks like the study drug but has no active ingredient.

All participants will be asked to take one capsule at the same time each day throughout the study.

This multi-center trial will be conducted in China. The overall time to participate in this study is up to 39 weeks. Participants will make 7 visits to the clinic, and will be contacted by telephone 5 to 10 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has endoscopically confirmed EE as defined by the LA Classification Grading System (A-D).

Exclusion Criteria:

1. Participant is required to take excluded medications, or it is anticipated that the participant will require treatment with at least 1 of the disallowed concomitant medications during the study evaluation period.
2. Has a hypersensitivity to any proton pump inhibitor (PPI) (including, but not limited to, lansoprazole, omeprazole, rabeprazole, pantoprazole, esomeprazole or ilaprazole), any component of dexlansoprazole, or antacid (example, magnesium trisilicate or similar antacid).
3. Had a history of cancer, (except basal cell carcinoma of the skin), that has not been in remission for at least 5 years prior to Screening.
4. Has a known history or any suspicious Barrett's esophagus with dysplastic changes seen during screening endoscopy.
5. Developed acute upper gastrointestinal bleeding, gastric ulcer (a mucosal defect with white coating) or duodenal ulcer (a mucosal defect with white coating), within 30 days before the start of the Screening Visit (with the possible inclusion of those with gastric or duodenal erosion). The participant requires chronic use (>12 doses per month) of non steroidal anti-inflammatory drugs (NSAIDs) including cyclooxygenase-2 (COX-2) NSAIDs within 30 days prior to the Screening Period and throughout the study.
6. Has comorbidities that could affect the esophagus (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal strictures); a history of radiotherapy or cryotherapy of the esophagus; and a history of corrosive or physiochemical injury (with the possible inclusion in the study of those with Schatzki's ring).
7. Has a history of surgical procedures that may affect the esophagus (example, fundoplication and mechanical dilatation for esophageal strictures) or a history of gastric or duodenal surgery other than endoscopic removal of benign polyps.
8. Participant is known to have the acquired immunodeficiency syndrome (AIDS) or hepatitis, including hepatitis virus carriers (that is, hepatitis B surface antigen HBs-antigen (HBsAg) positive or hepatitis C virus (HCV)-antibody positive).
9. Has current Zollinger-Ellison syndrome (gastric acid hyper secretion) or a history of gastric acid hypersecretion.
10. Participant is scheduled for surgery that requires hospitalization or requires surgical treatment during his/her participation in the study.
11. Has donated or lost >300 milliliter (mL) blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study drug.
12. Has a history of alcohol or drug abuse (defined as any illicit drug use), or drug addiction in the 12 months prior to Screening.
13. The participant with positive serology result of Helicobacter pylori (H. pylori) that needs eradication therapy during the study participation period as anticipated by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (25):
- China (25):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chong Qing
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Affilicated Hospital of Guilin Medical University, Haikou, Gui Lin
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Taihe Hospital, Shiyan, Hubei
  - Central Hospital of Wuhan, Wuhan, Hubei
  - Puai Hospital Of Wuhan City, Wuhan, Hubei
  - The Third Hospital of Changsha, Changsha, Hunan
  - Zhongda Hospital Southeast, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Wuxi, Jiangsu
  - Wuxi people's hospital, Wuxi, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Liaocheng Hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital,Sichuan University, Chengdu, Si Chuang
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- See also: Dexlansoprazole Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in China from 21 December 2016 to 06 November 2017.
Pre-assignment Details: Participants with erosive esophagitis (EE) were enrolled to receive: lansoprazole 30 milligram (mg) or dexlansoprazole 60 mg in Healing Period and dexlansoprazole 30 mg or Placebo in Maintenance Period. Study was terminated since compound was not expected to provide sufficient additional benefit to participants over currently available therapies.
Groups:
- Healing Period: Dexlansoprazole 60 mg: Dexlansoprazole 60 mg, capsules, orally, once daily for up to 8 weeks in the Healing Period.
- Maintenance Period: Placebo: Dexlansoprazole placebo-matching capsules, orally, once daily for up to 6 months in the Maintenance period. Participants who were healed at Week 8 entered the Maintenance Period.
- Maintenance Period: Dexlansoprazole 30 mg: Dexlansoprazole 30 mg, delayed-release capsules, orally, once daily for up to 6 months in the Maintenance period. Participants who were healed at Week 8 entered the Maintenance Period.
Period: Healing Period (up to Week 8)
Arm/Group | Healing Period: Lansoprazole 30 mg | Healing Period: Dexlansoprazole 60 mg | Maintenance Period: Placebo | Maintenance Period: Dexlansoprazole 30 mg
Started | 20 | 17 | 0 | 0
Completed | 19 | 16 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Maintenance Period (up to Month 6)
Arm/Group | Healing Period: Lansoprazole 30 mg | Healing Period: Dexlansoprazole 60 mg | Maintenance Period: Placebo | Maintenance Period: Dexlansoprazole 30 mg
Started | 0 | 0 | 8 | 8
Completed | 0 | 0 | 1 | 6
Not Completed | 0 | 0 | 7 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Relapse of EE | 0 | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set for the healing period (FAS-H) included all randomized participants who had documented EE at screening and had received at least 1 dose of study drug during the first 8 weeks of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healing Period: Lansoprazole 30 mg | Healing Period: Dexlansoprazole 60 mg | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (14.35) | 47.4 (11.03) | 48.4 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 17 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 20 | 17 | 37
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.28 (8.091) | 167.82 (8.346) | 166.99 (8.131)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 64.73 (10.002) | 69.44 (11.190) | 66.89 (10.683)
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 23.310 (2.2623) | 24.606 (3.5321) | 23.905 (2.9452)
BMI Categories [Count of Participants; unit: Participants]
  Less than (<) 25 kg/m^2 | 15 | 9 | 24
  25 to <30 kg/m^2 | 5 | 7 | 12
  Greater than or equal to (>=) 30 kg/m^2 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Healing Period: Percentage of Participants With Complete Healing of EE at Week 8
Description: Percentage of participants with complete healing of EE was assessed by endoscopy. EE was graded according to the Los Angeles (LA) classification of esophagitis grading system, based on the extent of visible mucosal breaks seen in the esophagus according to the following: Grade O (no mucosal breaks); Grade A (>=1 mucosal break no longer than 5 millimeter [mm] that does not extend between the tops of 2 mucosal folds); Grade B (>=1 mucosal break greater than [>] 5 mm that does not extend between the tops of 2 mucosal folds); Grade C (>=1 mucosal break that is continuous between the tops of 2 or more mucosal folds, but involves <75 percent (%) of the circumference); Grade D (>=1 mucosal break which involves >=75% of the circumference). Healing is defined as LA Grade O.
Time Frame: Week 8
Population: The FAS-H included all randomized participants who had documented EE at screening and had received at least 1 dose of study drug during the first 8 weeks of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Healing Period: Lansoprazole 30 mg | Healing Period: Dexlansoprazole 60 mg
Number analyzed (Participants) | 20 | 17
percentage of participants | 85.0 | 82.4
Statistical Analysis 1: Comparison: Healing Period: Lansoprazole 30 mg vs Healing Period: Dexlansoprazole 60 mg; Healing Period: Dexlansoprazole 60 mg versus Healing Period: Lansoprazole 30 mg; Test type: Non-Inferiority — Non-inferiority to lansoprazole if the lower bound of confidence interval (CI) for the treatment difference is greater than -10%; Difference in Percentage = -2.65, 95% CI 2-sided [-26.59 to 21.30]

2. Secondary Outcome: Maintenance Period: Percentage of Participants Who Maintained Complete Healing of EE at Month 6
Description: Percentage of participants with complete healing of EE was assessed by endoscopy. EE was graded according to the LA classification of esophagitis grading system, based on the extent of visible mucosal breaks seen in the esophagus according to the following: Grade O (no mucosal breaks); Grade A (>=1 mucosal break no longer than 5 mm that does not extend between the tops of 2 mucosal folds); Grade B (>=1 mucosal break >5 mm that does not extend between the tops of 2 mucosal folds); Grade C (>=1 mucosal break that is continuous between the tops of 2 or more mucosal folds, but involves <75% of the circumference); Grade D (>=1 mucosal break which involves >=75% of the circumference). Healing is defined as LA Grade O.
Time Frame: Month 6
Population: The full analysis set for the maintenance period (FAS-M) included all participants with healed EE by week 8 who were randomized and received at least 1 dose of study drug during 6 months of maintenance treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Period: Placebo | Maintenance Period: Dexlansoprazole 30 mg
Number analyzed (Participants) | 8 | 8
percentage of participants | 0 | 25

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 5 to 10 days (Day 190) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Healing Period: Lansoprazole 30 mg | Healing Period: Dexlansoprazole 60 mg | Maintenance Period: Placebo | Maintenance Period: Dexlansoprazole 30 mg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 15/20 | 7/17 | 1/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healing Period: Lansoprazole 30 mg (N=20) | Healing Period: Dexlansoprazole 60 mg (N=17) | Maintenance Period: Placebo (N=8) | Maintenance Period: Dexlansoprazole 30 mg (N=8)
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT02873702/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT02873702/SAP_001.pdf